CLINICAL TRIAL: NCT05525585
Title: Early Human Milk Fortification After Early, Exclusive, Enteral Nutrition in Very Preterm Infants: a Randomized Clinical Trial
Brief Title: Early Human Milk Fortification After Early, Exclusive, Enteral Nutrition in Very Preterm Infants
Acronym: ENACT+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, Ariel A. Salas, Associate Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 300009921; 000538159 (Other Grant/Funding Number: Mead Johnson Nutrition)
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Prematurity; Light-For-Dates; Enteral Feeding Intolerance
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early human milk fortification (HMF) group (Experimental): A human milk fortifier will be added to the feeds between days 4 to 7, after a total feeding volume greater than 120 ml/kg/day is achieved.
  Interventions: Dietary Supplement: Early HMF
- Delayed human milk fortification (HMF) group (Active Comparator): A human milk fortifier will be added to the feeds between days 10 to 14, after a total feeding volume greater than 120 ml/kg/day is achieved.
  Interventions: Dietary Supplement: Delayed HMF

INTERVENTIONS:
Dietary Supplement: Early HMF — Mom's milk or donor milk will be fortified between postnatal day 4 and 7
  Arms: Early human milk fortification (HMF) group
Dietary Supplement: Delayed HMF — Mom's milk or donor milk will be fortified between postnatal day 10 and 14
  Arms: Delayed human milk fortification (HMF) group

SUMMARY:
In this proposed clinical trial, the investigators will randomize 80 very preterm (VPT) infants to receive either early (between day 4 and 7) or delayed (between day 10 and 14) fortification and determine if providing early protein supplementation through early fortification results in higher FFM-for-age z scores and more diversity in the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 29 to 33 weeks of gestation
* Birth weight < 1800 g
* Postnatal age < 96 hours

Exclusion Criteria:

* Small for gestational age (<5th percentile)
* Major congenital/chromosomal anomalies
* Terminal illness needing withhold or limit support

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Fat-free mass(FFM)-for-age Z-score | Postnatal day 14 to 21
  Estimated by air displacement plethysmography

SECONDARY OUTCOMES:
Fecal microbiome composition | Birth to 36 weeks postmenstrual age
  Determined by 16S RNA sequencing of bacteria in stool samples
Growth - Weight | Birth to 36 weeks postmenstrual age or hospital discharge
  Measured weekly in grams and z scores as part of routine care
Growth - Length | Birth to 36 weeks postmenstrual age or hospital discharge
  Measured weekly in cm and z scores as part of routine care
Growth - Head circumference | Birth to 36 weeks postmenstrual age or hospital discharge
  Measured weekly in cm and z scores as part of routine care
Growth rate | Birth to 36 weeks postmenstrual age or hospital discharge
  Weight gain in g/kg/day
Number of participants with postnatal growth faltering | Birth to 36 weeks postmenstrual age or hospital discharge
  Diagnosis of growth faltering (decline in weight-for-age z score from birth to 36 weeks postmenstrual age greater than 1.2
Number of participants with diagnosis of necrotizing enterocolitis | Birth to 60 days or discharge
  Diagnosis of necrotizing enterocolitis stage 2 or 3
Number of participants with diagnosis of intestinal perforation | Birth to 10 days
  Diagnosis of intestinal perforation
Death | Birth to 60 days
  Death prior to postnatal day 60
Duration of hospital stay in days | Birth to 60 days or discharge, whichever occurs first
  From day of admission to day of hospital discharge to home

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A. Salas, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Salas AA, Gunawan E, Jeffcoat S, Nguyen K. Early full enteral nutrition with fortified milk in very preterm infants: a randomized clinical trial. Am J Clin Nutr. 2025 May;121(5):1117-1123. doi: 10.1016/j.ajcnut.2025.02.019. Epub 2025 Feb 21. PMID 39986385